CLINICAL TRIAL: NCT04972162
Title: Web App Fitting Strategy Validation NSR Device Study
Brief Title: Fitting Strategy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WSAUD A/S (Industry)
Collaborators: University of South Dakota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D00232675
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The masking only done at the final visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Web-App-fitted Hearing Aid, Then Standard-of-care fitted Hearing Aid (Experimental): Patients self-fitted the web-app-fitted hearing aids and wore them in a home-trial for 14 days. After a washout period of 5 days, they were fitted by a hearing care professional with the Standard-of-care fitted hearing aids and wore those in a home-trial for 14 days.
  Interventions: Device: Web App Strategy Fitting; Device: Standard-of-care Fitting
- Standard-of-care-fitted Hearing Aid, Then Web-App-fitted hearing Aid (Experimental): Patients were fitted by a hearing care professional with the Standard-of-care fitted hearing aids and wore them in a home-trial for 14 days. After a washout period of 5 days, they self-fitted the web-app-fitted hearing aids and wore those in a home-trial for 14 days.
  Interventions: Device: Web App Strategy Fitting; Device: Standard-of-care Fitting

INTERVENTIONS:
Device: Web App Strategy Fitting — Web App Strategy fitting of hearing aids
Device: Standard-of-care Fitting — Standard-of-care fitting of hearing aids

SUMMARY:
To be conducted with adult participants with mild-to-moderate hearing loss to validate the effectiveness of the Web App fitting strategy. Validation measures participant's perceived hearing aid benefit when using the Web App fitted hearing aids and when using standard-of-care fitted hearing aids.

DETAILED DESCRIPTION:
A prospective, randomized controlled, adaptive design, non-inferiority, pre-market and NSR device study. Completed in 26 adult subjects with mild-to-moderate hearing loss to validate the effectiveness of a Web App fitting strategy. Validation measured subject´s perceived hearing aid benefit when using the Web App fitted hearing aids and when using standard-of-care fitted hearing aids.

The adaptive study design began with a cross-over design of the first 12 subjects. At the interim analysis, the possibility of an interaction effect was evaluated as a nuisance parameter. In the absence of an interaction effect, the study was completed in cross-over design.

The standard-of-care fitted hearing aids were fitted to National Acoustic Laboratories Nonlinear Version 2 (NAL-NL2) prescriptive targets, verified by probe-mic real-ear measures (REM). The null hypothesis (H0) was that subject´s perceived hearing aids benefit using Web App fitted hearing aids is inferior to perceived benefit using standard-of-care fitted hearing aids, and the alternative hypothesis (Ha) was that subject´s perceived hearing aids benefit using Web App fitted hearing aids is non-inferior to that using standard-of-care fitted hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older,
* Self-perceived mild to moderate hearing impairment,
* Signed informed consent form (ICF),
* Fluent in English listening and reading comprehension,
* With or without prior experience with hearing aids. At least four subjects and maximum 30% of the total number of subjects enrolled in this study will have prior hearing aid experience.
* Measured audiogram with at least four of the test frequencies 500 Hz, 1000 Hz, 2000 Hz, 3000 Hz, and 4000 Hz within fitting range of Web App fitted hearing aid

Exclusion Criteria:

* Hearing aids do not fit into the person's ears with any of the offered silicone 'Click Sleeves' instant ear tips.
* Abnormal conditions:

  * Severe hearing loss or deafness in at least one ear.
  * A steep decline in hearing ability within the last 90 days in one or both ears.
  * Active discharge within the last 90 days.
  * Dizziness.
  * A visible deformity of the ear.
  * Pain, or discomfort in the ear, or significant ear wax accumulation.
  * Audiometric air-bone gap equal to or greater than 15 decibels at 500 hertz Hz, 1,000 Hz, and 2,000 Hz.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Jorgensen, Principal Investigator — University of South Dakota
Locations (1):
- University of South Dakota, USD Speech and Hearing Clinic, Vermillion, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard-of-care Fitted Hearing Aid, Then Web-App-fitted Hearing Aid: Patients were fitted by a hearing care professional with the Standard-of-care fitted hearing aids and wore them in a home-trial for 14 days. After a washout period of 5 days, they self-fitted the web-app-fitted hearing aids and wore those in a home-trial for 14 days.
Period: First Intervention (14 Days)
Arm/Group | Web-App-fitted Hearing Aid, Then Standard-of-care Fitted Hearing Aid | Standard-of-care Fitted Hearing Aid, Then Web-App-fitted Hearing Aid
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout Period (5 Days)
Arm/Group | Web-App-fitted Hearing Aid, Then Standard-of-care Fitted Hearing Aid | Standard-of-care Fitted Hearing Aid, Then Web-App-fitted Hearing Aid
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (14 Days)
Arm/Group | Web-App-fitted Hearing Aid, Then Standard-of-care Fitted Hearing Aid | Standard-of-care Fitted Hearing Aid, Then Web-App-fitted Hearing Aid
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Baseline measures are only given for the total group of study participants because of the cross-over design (all participants took part in both arms)
Arm/Group | Study Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Self-perceived hearing loss [Count of Participants; unit: Participants] | 28
Prior experience with hearing aids [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The APHAB consists of 24 questions across 4 subscales: Ease of Communication (EC), Background Noise (BN), Reverberation (RV), and Aversiveness (AV), assessing hearing difficulties in daily situations reported as percentage of problems (0-100%, 100% = highest number of problems). It evaluates hearing aid (HA) benefit by subtracting the reported % of problems with HA from without HA, yielding scores from 0 (no benefit) to 100 (maximum benefit) in each subscale. The study focuses on the communication subscales (EC, BN, RV) and calculates benefit score differences for each subscale after using A) Web-App-fitted and B) standard-of-care-fitted HAs. The difference-of-benefit scores are compared to non-inferiority margins from Cox&Alexander (Ear&Hearing 1995). Differences-in-benefit scores range from -100 to 100, with negative scores indicating greater benefit with Web-App-fitted HAs, 0 indicating identical benefit and higher scores indicating greater benefit with standard-of-care fitting.
Time Frame: 14-17 Days hearing aid wearing time per fitting type
Population: All participants who completed the study visits were included in the efficacy analysis. The intention to treat (ITT) population includes 2 subjects who withdrew from study. It was concluded that their primary endpoint data was missing for cause and their APHAB benefit scores (change from baseline) was imputed as 0 for each subscale
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Web-App-fitted Hearing Aids: Participants who wore the web-app-fitted hearing aids either the first or last 2 weeks of the study
- Standard-of-care-fitted Hearing Aids: Participants who wore the standard-of-care-fitted hearing aids either the first or last 2 weeks of the study
Arm/Group | Web-App-fitted Hearing Aids | Standard-of-care-fitted Hearing Aids
Number analyzed (Participants) | 26 | 26
score on a scale
  Benefit Ease of Communication | 12.7 (19.09) | 13.18 (13.60)
  Benefit Background Noise | 11.17 (22.98) | 12.22 (19.94)
  Benefit Reverberant Room | 11.43 (22.32) | 12.49 (16.76)
Statistical Analysis 1: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Check for interaction effect for Ease of Communication Subscale (EC) The statistical analysis method was a repeated-measures ANOVA in which: * order is a "between-subjects" effect - i.e., each subject has just one order * treatment is a "within-subjects" effect - i.e., each subjects has both treatments because of the cross-over design * the interaction term treatment x order is a "within-subjects" effect. The rm-ANOVAs generates a nuisance p-value: that of the interaction effect; Test type: Other — The rm-ANOVA model fitted for the primary analysis was run to confirm if there is a significant interaction for treatment and order. This confirmation of the absence of an interaction effect is needed to validate the pooling of the two periods of Web-App treatment and the two periods of Standard-of-Care treatment, respectively; p = 0.38, ANOVA — p<0.05 would show that there is an interaction effect i.e. results would differ depending on the order in which the participants wore the hearing aids
Statistical Analysis 2: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Check for interaction effect for Background Noise Subscale (BN) The statistical analysis method was a repeated-measures ANOVA in which: * order is a "between-subjects" effect - i.e., each subject has just one order * treatment is a "within-subjects" effect - i.e., each subjects has both treatments because of the cross-over design * the interaction term treatment x order is a "within-subjects" effect. The rm-ANOVAs generates a nuisance p-value: that of the interaction effect; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.79, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Check for interaction effect for Reverberant Room Subscale (RV) The statistical analysis method was a repeated-measures ANOVA in which: * order is a "between-subjects" effect - i.e., each subject has just one order * treatment is a "within-subjects" effect - i.e., each subjects has both treatments because of the cross-over design * the interaction term treatment x order is a "within-subjects" effect. The rm-ANOVAs generates a nuisance p-value: that of the interaction effect; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.51, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Results for Ease of Communication Subscale. Null hypothesis: benefit(standard-of-care fit) - benefit(web-app-fit) < noninferiority margin for all subscales. Each subscale was analyzed using an rm-ANOVA in which the repeated factors are order & treatment; no between-group factors. Interaction term was order x treatment. ITT population includes 2 subjects who withdrew. It was concluded that their primary endpoint data was missing for cause and their APHAB benefit scores were imputed as 0; Test type: Non-Inferiority — Non-inferiority tests compared the subject´s perceived hearing aid benefit when the hearing aid was standard-of-care fitted compared to Web-App fitted by the subject. The non-inferiority margins are the minimum clinically important differences on each of the 3 communication benefit subscales as described by Cox & Alexander (Ear and Hearing 1995;16;176-186). These literature values are as follows: Ease of Communication (EC): 26, Background Noise (BN): 27, Reverberant Room (RV): 28; p < 0.0001, ANOVA — Threshold for statistical significance was p =0.05. p-value was calculated using the estimated difference of benefits, calculating a new t-statistic by subtracting the applicable non-inf. margin from the difference and dividing by standard error; repeated measures ANOVA where factors are order and treatment is device with patient as a random effect. Added interaction term of treatment and order; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-4.3 to 5.2] — Difference calculated as benefit(standard-of-care fit) - benefit(web-app-fit)
Statistical Analysis 5: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Results for Background Noise Subscale. Null hypothesis: benefit(standard-of-care fit) - benefit(web-app-fit) < noninferiority margin for all subscales. Each subscale was analyzed using an rm-ANOVA in which the repeated factors are order & treatment; no between-group factors. Interaction term was order x treatment. ITT population includes 2 subjects who withdrew. It was concluded that their primary endpoint data was missing for cause and their APHAB benefit scores were imputed as 0; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-5.3 to 7.2] — Difference calculated as benefit(standard-of-care fit) - benefit(web-app-fit)
Statistical Analysis 6: Comparison: Web-App-fitted Hearing Aids vs Standard-of-care-fitted Hearing Aids; Results for Reverberant Room Subscale. Null hypothesis: benefit(standard-of-care fit) - benefit(web-app-fit) < noninferiority margin for all subscales. Each subscale was analyzed using an rm-ANOVA in which the repeated factors are order & treatment; no between-group factors. Interaction term was order x treatment. ITT population includes 2 subjects who withdrew. It was concluded that their primary endpoint data was missing for cause and their APHAB benefit scores were imputed as 0; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [-4.6 to 6.5] — Difference calculated as benefit(standard-of-care fit) - benefit(web-app-fit)

ADVERSE EVENTS:
Time Frame: through study completion, starting with visit 1 and ending with visit 3 after the second field test. Approximately 5 weeks for each patient.
Groups:
- Web App Fitted Hearing Aids: Web App fitted hearing aids will be worn by subject for 14 days.
  Web App Strategy Fitting: Web App Strategy fitting of hearing aids
- Standard-of-care Fitted Hearing Aids: Standard-of-care fitted hearing aids will be worn by subject for 14 days.
  Standard-of-care Fitting: Standard-of-care fitting of hearing aids
Arm/Group | Web App Fitted Hearing Aids | Standard-of-care Fitted Hearing Aids
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT04972162/Prot_SAP_000.pdf